CLINICAL TRIAL: NCT06403202
Title: Prognostic Performance of a Chemogram in Patients With Intermediate-grade Superficial Bladder Cancer and Invasive Bladder Cancer: Proof of Concept.
Brief Title: Prognostic Performance of a Chemogram in Patients With Bladder Cancer.
Acronym: CHEMOGRAM
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC-P0095
Record Dates: First submitted 2024-04-19; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Urinary Bladder Neoplasms; Chemogram
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate chemogram in patients with intermediate-grade superficial bladder cancer and patients with infiltrating bladder cancer, who are likely to be treated according to the standard procedure. This project is based on the premise that treatments - notably chemotherapy - are standard, but that each cancer is unique. It is therefore necessary to personalize the treatment for each patient, while at the same time proposing an approach that is economically bearable for the healthcare system. For both types of bladder tumor, chemotherapy is used either as an alternative to immunotherapy, or as an adjuvant to surgery. Its use is therefore based on its effectiveness in reducing post-treatment recurrence.

DETAILED DESCRIPTION:
The project is based on the premise that treatments - particularly chemotherapy - are standard, but that each cancer is unique. It is therefore necessary to personalize treatment for each patient, while proposing an approach that is economically viable for our healthcare system. The chemogram is inspired by the principle of antibiograms, since it tests, for a given patient and in conjunction with oncologists, different chemotherapeutic or targeted treatment options based on clinical and anatomopathological data. These tests are carried out in vitro in academic research laboratories.

With this study, its proposed a "proof of concept" for the clinical use of chemograms in patients with superficial or infiltrating bladder cancer. The use of chemograms will have no impact whatsoever on the patient's treatment, which will be administered according to standard practice. Nevertheless, this study may help determine whether chemograms can detect tumor sensitivity to certain anti-cancer treatments.

In the years to come, the aim of this research work is to be able to guide the therapeutic management of patients whose tumours are resistant to the treatment envisaged (tumours with intrinsic resistance to treatment). This will avoid unnecessary treatments for the patient, often with very serious side effects.

For these two types of bladder tumour, the use of a chemogram to detect the tumour's chemosensitivity would make treatment more effective and rapid.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with suspected bladder cancer likely to be treated with chemotherapy
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Insufficient tumor volume
* Patient under guardianship
* Pregnant or breast-feeding women
* Patient opposed to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate-grade superficial bladder cancer and invasive bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Chemogram sensitivity | 12 months
  The relevance of the chemogram to the patient's response to treatment will be assessed by calculating sensitivities, the gold standard being the proven response of patients with infiltrative bladder tumors to treatment.
Chemogram specificity | 12 months
  The relevance of the chemogram to the patient's response to treatment will be assessed by calculating specificity, the gold standard being the proven response of patients with infiltrative bladder tumors to treatment.
Positive predictive value | 12 months
  The relevance of the chemogram to the patient's response to treatment will be assessed by calculating positive predictive value, the gold standard being the proven response of patients with infiltrative bladder tumors to treatment.
Negative predictive value | 12 months
  The relevance of the chemogram to the patient's response to treatment will be assessed by calculating negative predictive value, the gold standard being the proven response of patients with infiltrative bladder tumors to treatment.

SECONDARY OUTCOMES:
Proteomic analysis | 12 months
  Proteomic analysis will detect various endogenous compounds: metabolites, lipids, peptides and proteins. Protein profiles (chemo-sensitive cancer, chemo-insensitive cancer, non-cancer) can be identified.
  and/or transcriptomic
Transcriptomic analysis | 12 months
  and/or transcriptomic

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Bonnal, Principal Investigator — GHICL
Locations (1):
- Hôpital St Philibert, Lomme, France